CLINICAL TRIAL: NCT07204665
Title: European Study in Colon Obstruction
Brief Title: This Study Has Been Designed to Support the Working Hypothesis That Emergency Surgery in a Colon Obstruction Neoplasm is Better Than Stent Bridge Due to Better Oncological Outcomes, Analyzing the Importance of ERAS Programs in Emergency Colon Obstruction Surgery.
Acronym: EUCOBS
Status: Enrolling by invitation | Type: Observational
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Jose-M Ramirez, Full Professor, Universidad de Zaragoza
Other Study IDs: EUCOBS
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Colon Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urgent: Patients with urgent surgery
- Elective: Patients with elective surgery

SUMMARY:
This study has been designed to support the working hypothesis that emergency surgery in a colon obstruction neoplasm is better than stent bridge due to better oncological outcomes. The primary objective is to analyse the importance of ERAS program implementation in emergency colon obstruction surgery

ELIGIBILITY:
Inclusion Criteria

* All adult patients (aged >18 years) with a diagnosis of Malignant obstruction colorectal cancer. Informed consent will be obtained from all subjects who will participate in the study voluntarily.
* ASA I, II and III
* No more than 5 days from symptoms onset.
* Absence of proximal colon severe dilatation( no more than 8 centimeters), severe malnutrition.
* No Inmunocompromised patients
* Patients suffer from segmentary colectomy, with or without anastomosis with o witjhout lateral ileostomy
* Patients suffer from Hartmann procedure.

Exclusion criteria:

* Patient refusal.
* Patients under 18 years of age.
* ASA IV
* Stent placement
* ICU stay more than 2 days
* Peritonitis
* Out of protocol if patient would need total parenteral nutrition(NPT) during postoperative or Clavien-Dindo more or equal than II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged >18 years) with a diagnosis of Malignant obstruction colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | From enrollment to 90 days
  The primary objective is to analyse the importance of ERAS program implementation in emergency colon obstruction surgery

SECONDARY OUTCOMES:
1 year survival analysis | 360 days after surgery
  1 year survival analysis
Overall survival | 365 days after surgery
  Overall survival
disease-related survival | 365 days after surgery
  disease-related survival
disease-free survival | 365 days after surgery
  disease-free survival
Relationship between stent bridge and colon perforation | 60 days after stent placement
  Relationship between stent bridge and colon perforation

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Urduliz, Bilbao, Vizcaya, Spain